CLINICAL TRIAL: NCT07005960
Title: The Effect of Art Therapy on Anxiety and Psychological Resilience in Patients Undergoing Hemodialysis Treatment
Brief Title: The Application of Art Therapy to Patients Undergoing Hemodialysis Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EMİNE İNAL (Other)
Responsible Party: Sponsor-Investigator, EMİNE İNAL, Principal İnvestigator, Cyprus Aydin University
Organization: Cyprus Aydin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CAU-LEAE-HEM-Eİ-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Psychological Well-Being; Hemodialysis
Keywords: Art therapy; Art therapy applied to hemodialysis patients; Anxiety and Psychological Well-Being
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: Two groups, experimental group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: A total of 35 participants each for the experimental and for control groups will be randomly selected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art therapy experimental group (Active Comparator): Patients in the experimental group will be administered the Volunteer Information and Consent Form, the Patient Information Form, the Brief Resilience Scale, and the State-Trait Anxiety Inventory prior to the intervention.
  Interventions: Other: Art Therapy for Anxiety in Hemodialysis Patients; Other: Art Therapy for Resilience in Hemodialysis Patients
- Art therapy control group (Active Comparator): For the control group (35 participants), during the first week, without any intervention beyond standard clinical procedures, participants will complete the Volunteer Information and Consent Form, the Patient Information Form, the Brief Resilience Scale, and the State-Trait Anxiety Inventory. This process will be repeated in the fourth week. One month later, the same scales will be administered again without any intervention.
  Interventions: Other: Art Therapy for Anxiety in Hemodialysis Patients; Other: Art Therapy for Resilience in Hemodialysis Patients

INTERVENTIONS:
Other: Art Therapy for Anxiety in Hemodialysis Patients — Patients in the experimental group will be administered the Volunteer Information and Consent Form, the Patient Information Form, and the State-Trait Anxiety Inventory prior to the intervention.
  Then, for four weeks, the experimental group will participate in art therapy sessions involving drawing and painting for approximately 30 minutes, twice a week. In the first week, patients will be asked to paint a given picture. In the second week, they will be given a different picture to paint. In the third week, they will be asked to draw and paint a picture of their choice. In the fourth week, they will again be asked to draw and paint a picture of their choice. At the end of the fourth week, the scales will be completed again.
  After this, there will be a one-month break from art therapy, during which no intervention will be conducted. At the end of this month, the same scales will be administered again to the experimental group.
Other: Art Therapy for Resilience in Hemodialysis Patients — Patients in the experimental group will be administered the Volunteer Information and Consent Form, the Patient Information Form, the Brief Resilience Scale, prior to the intervention.
  Then, for four weeks, the experimental group will participate in art therapy sessions involving drawing and painting for approximately 30 minutes, twice a week. In the first week, patients will be asked to paint a given picture. In the second week, they will be given a different picture to paint. In the third week, they will be asked to draw and paint a picture of their choice. In the fourth week, they will again be asked to draw and paint a picture of their choice. At the end of the fourth week, the scales will be completed again.
  After this, there will be a one-month break from art therapy, during which no intervention will be conducted. At the end of this month, the same scales will be administered again to the experimental group.

SUMMARY:
Purpose of the Study: This study aims to investigate the effect of art therapy on anxiety and psychological resilience levels in Chronic kidney disease(CKD) patients undergoing hemodialysis patients.

Hemodialysis patients undergo long-term treatment, often experiencing psychological issues such as anxiety and depression, which significantly reduce their quality of life. Among non-pharmacological approaches to alleviate these symptoms, art therapy has gained increasing attention. Art therapy helps patients shift their focus away from their illness, fosters self-confidence, reduces anxiety, and promotes relaxation .

DETAILED DESCRIPTION:
Preliminary Implementation of the Study Implementation of the Research During the data collection phase of the study, the researcher will explain the purpose of the study to patients who meet the inclusion criteria, provide necessary information, and obtain both verbal and written informed consent. After the information and consent process, all data in the "Personal Information Form" related to the patient will be filled out by the researcher.

Patients will be divided into two groups: the experimental group (35 participants) and the control group (35 participants). Patients in the experimental group will be administered the Volunteer Information and Consent Form, the Patient Information Form, the Brief Resilience Scale, and the State-Trait Anxiety Inventory prior to the intervention.

Then, for four weeks, the experimental group will participate in art therapy sessions involving drawing and painting for approximately 30 minutes, twice a week. In the first week, patients will be asked to paint a given picture. In the second week, they will be given a different picture to paint. In the third week, they will be asked to draw and paint a picture of their choice. In the fourth week, they will again be asked to draw and paint a picture of their choice. At the end of the fourth week, the scales will be completed again. By this point, each patient will have painted four given pictures and drawn and painted four of their own.

After this, there will be a one-month break from art therapy, during which no intervention will be conducted. At the end of this month, the same scales will be administered again to the experimental group.

For the control group (35 participants), during the first week, without any intervention beyond standard clinical procedures, participants will complete the Volunteer Information and Consent Form, the Patient Information Form, the Brief Resilience Scale, and the State-Trait Anxiety Inventory. This process will be repeated in the fourth week. One month later, the same scales will be administered again without any intervention.

ELIGIBILITY:
Inclusion Criteria:

Undergoing hemodialysis for at least 6 months,

Willing to participate in the study,

Aged between 18 and 65 years,

No communication disorders,

No infectious diseases.

Exclusion Criteria:

Sensory impairments (vision or hearing loss),

Not willing to participate in the study,

Having an infectious disease.

Independent and Dependent Variables:

Independent Variable: Art therapy. Dependent Variables: Scores from the Brief Resilience Scale and State-Trait Anxiety Inventory (STAI 1-STAI 2).

Control Variables: Participants' sociodemographic characteristics.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
State And Trait Anxiety Scale | 2 months
  Measuring the change in Anxiety Levels through art therapy in patients undergoing hemodialysis treatment.
Brief Psychological Resilience Scale | 2 months
  Measuring the change in Psychological Resilience Levels through art therapy in patients undergoing hemodialysis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Olca POLAT, Study Director — sibelolca@aydın.edu.tr
Locations (1):
- Çeşme Alper Çizgenakat State Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No